CLINICAL TRIAL: NCT01282515
Title: A Study of Topical Hexaminolevulinate (HAL) Photodynamic Therapy (PDT) and a Phase III Comparative Treatment Study of HAL PDT in Female Genital Erosive Lichen Planus (GELP)
Brief Title: Treatment of Female Genital Erosive Lichen Planus(GELP) With Hexaminolevulinate PDT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Photocure (Industry)
Responsible Party: Principal Investigator, Anne Lise Helgesen, consultant dermatologist, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALH ELP 2/10
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Genital Lichen Planus
MeSH Terms: interventions — Clobetasol; Ointments; 5-aminolevulinic acid hexyl ester

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ELP active (Experimental): one PDT treatment with 2 ml hexaminolevulinate 6 mg/ml gel
  Interventions: Drug: hexaminolevulinate
- topical steroids (Active Comparator): treatment with clobetasol propionate 0.05% ointment used daily for 6 weeks
  Interventions: Drug: clobetasol propionate 0,05% ointment

INTERVENTIONS:
Drug: clobetasol propionate 0,05% ointment — continuously daily treatment for 6 weeks
  Other Names: Dermovate 0.05% ointment
  Arms: topical steroids
Drug: hexaminolevulinate — one PDT treatment
  Arms: ELP active

SUMMARY:
To compare the effect and side effects of photodynamic treatment and traditional topical steroid treatment in female genital erosive lichen planus

DETAILED DESCRIPTION:
To assess the feasibility, efficacy and safety of hexyl 5-aminolevulinate-hydrocloride (HAL)-PDT in GELP in women.

ELIGIBILITY:
Inclusion Criteria:

Women with symptomatically genital ELP, clinically verified by at least one doctor attended to the Vulva clinic.

Untreated for ELP for at least 4 weeks. Written Informed Consent signed Age 18 or above

Exclusion Criteria:

Current pelvic inflammatory disease, genital malignancy, or gynecological infection.

Known or suspected porphyria

Known allergy to hexaminolevulinate or similar compounds (e.g. hexaminolevulinate or aminolevulinic acid) Pregnancy and lactation Participation in other clinical study either concurrently or within the last 30 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Percentage change of GELP score and/or VAS score 6 weeks after start of treatment. | 6 weeks

SECONDARY OUTCOMES:
Percentage change of GELP score and/or VAS score 6 months after start of treatment. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: anne lise helgesen, md, Principal Investigator — research fellow
Locations (1):
- Rikshospitalet, OsloUniversity hospital, Oslo, Norway